CLINICAL TRIAL: NCT07070531
Title: Feasibility and Clinical Utility Study of the Unified Protocol for Group Treatment of Emotional Disorders in Penitentiary Facilities
Brief Title: Unified Protocol in Penitentiary Facilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Óscar Peris Baquero, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPES/PU-CP/2025
Record Dates: First submitted 2025-04-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Depression Disorders; Anxiety; Mood Disorders; Emotional Disorder
Keywords: Unified Protocol; Transdiagnostic Intervention; Incarcerated Population; Correctional Facilities; Group Therapy; Cognitive-behavioral Therapy; Emotional Disorders
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: The recruitment process for this study will be conducted within the participating correctional facilities: Brians 1, Brians 2, Quatre Camins, and Lledoners (Barcelona). Inmates who are evaluated in the specialized Mental Health care service at the correctional facility and who have at least one diagnosis of a mental health disorder (TE) will be offered the opportunity to participate.
  The selection process will be based on the clinical evaluation carried out by the mental health professionals, who will inform the inmates about the possibility of participating in the study and offer them the chance to join, provided they meet the inclusion criteria and give their informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unified Protocol in group format (Experimental): Participants will receive the intervention of the Unified Protocol (UP) in a group format, consisting of 12 sessions, one per week, each lasting 1 hour. Each session includes a review of previous content, resolution of doubts, and development of new material from one of eight modules. The program covers motivation for change, goal setting, understanding the adaptive function of emotions, emotional awareness and mindfulness, cognitive flexibility, problem solving, and addressing emotion-driven behaviors. Exposure to emotional and interoceptive experiences is introduced in later sessions. Follow-up sessions at 1, 3, and 6 months review progress, reinforce learning, identify risk signals, and promote relapse prevention and long-term well-being.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol (UP) is a transdiagnostic, emotion-focused cognitive-behavioral treatment designed to address a range of emotional disorders, including anxiety, depression, and related conditions. It targets core mechanisms such as emotional avoidance, cognitive rigidity, and maladaptive emotion regulation strategies. The UP consists of structured modules focused on increasing emotional awareness, cognitive flexibility, and exposure to emotionally evocative situations. By addressing common underlying processes across disorders, the UP enhances treatment efficiency and applicability in both individual and group formats. Its flexibility makes it suitable for diverse populations and settings, including community and clinical contexts.

SUMMARY:
Emotional disorders (EDs), which include anxiety disorders, unipolar mood disorders, and other related conditions, exhibit a high prevalence within prison populations, significantly exceeding that of the general population. Despite the high incidence of these disorders, the resources available for their treatment in correctional facilities are limited. The shortage of both human and material resources hinders inmates' access to quality mental health care.

In this context, the Unified Protocol (UP) for the transdiagnostic treatment of emotional disorders, a transdiagnostic intervention grounded in Cognitive Behavioral Therapy, has demonstrated effectiveness in addressing a variety of psychological problems across different contexts. It has also proven to be cost-effective, particularly when delivered in a group format. Therefore, implementing the UP in group format within correctional settings could represent a viable strategy to optimize limited resources and provide accessible and effective treatment to a larger number of inmates.

The primary objective of this pilot study is to evaluate the feasibility and clinical utility of the UP for the treatment of emotional disorders in prison environments. To this end, the UP will be delivered to approximately 25 participants, organized into groups of six to eight individuals, each receiving 12 weekly sessions lasting one hour. Follow-up assessments will be conducted at one, three, and six months after the intervention.

A mixed-methods approach will be employed to analyze the results, combining quantitative analyses to assess changes in emotional symptomatology and qualitative analyses to explore participant satisfaction and therapist acceptance. It is expected that participants will experience statistically significant improvements in emotional symptoms and that these improvements will be sustained over time, up to the six-month follow-up. It is also anticipated that participants will report a high level of satisfaction with the treatment. Furthermore, therapists are expected to evaluate the intervention positively and to identify potential barriers to its implementation.

The results of this pilot study will contribute to improving the feasibility and clinical utility of the UP in correctional settings, while also laying the groundwork for a future randomized controlled trial involving a larger number of facilities, participants, and therapists.

DETAILED DESCRIPTION:
Prevalence of Mental Disorders in the Prison Population

According to the World Health Organization, mental disorders are the most prevalent health condition in European penitentiary institutions, affecting 32.8% of the incarcerated population, with incidence rates continuing to rise. This trend is corroborated by numerous studies that have long highlighted the high prevalence of mental disorders among inmates, significantly surpassing rates observed in the general population. For instance, common mental disorders (e.g., anxiety and mood disorders) are reported to be twice as prevalent, while severe mental disorders (e.g., personality or psychotic disorders) are up to four times more prevalent among the incarcerated population.

In Spain, the 2022 Survey on Health and Drug Use in the Inmate Population revealed that 42.3% of incarcerated women and 34.3% of incarcerated men have been diagnosed with a psychological disorder at some point in their lives. The study found prevalence rates of 18% for depression, 9.3% for personality disorders, and 5.6% for bipolar disorder. Similar results have been reported in other studies, where 14% of diagnoses among inmates were related to mood and/or anxiety disorders, with 80% of cases showing comorbidity with more than one diagnosis.

Conceptualization of Emotional Disorders and Emotion Dysregulation

Despite the diversity of disorders encompassed by anxiety and mood disorders and their differing clinical manifestations, scientific literature supports their grouping under a single category termed Emotional Disorders (EDs), which includes anxiety disorders, unipolar mood disorders, trauma- and stressor-related disorders, and obsessive-compulsive and related disorders. It has been suggested that these disorders share common etiological and maintenance mechanisms, such as neuroticism-defined as the trait tendency to experience frequent and intense negative emotions along with the perception of the world as dangerous/unpredictable -low extraversion, described as the tendency to engage with the environment with energy, joy, sociability, and confidence, and difficulties in emotion regulation, understood as the process by which an individual can influence the emotions they experience, how they experience them, and how and when they express them. Scientific evidence indicates that individuals with EDs exhibit deficits in emotion regulation and tend to engage in maladaptive emotion regulation behaviors, such as avoiding places, situations, sensations, or thoughts that are unpleasant, aiming to reduce emotional distress. While this may be effective in the short term by decreasing emotional discomfort, in the medium and long term, it not only fails to resolve the problem but also exacerbates and perpetuates it over time.

Mental Health Care in Spanish Prisons

Despite the high prevalence of mental disorders in this context, penitentiary centers have limited human and material resources. Specifically, in 2020, the estimated ratio of prison doctors per 1,000 inmates in Spain was 5.2, below the European average of 8.0 doctors per 1,000 inmates, according to WHO data. Similarly, the ratios of psychology or psychiatry professionals in penitentiary centers fall below international recommendations, with estimated ratios in 2020 of 0.8 psychiatric specialists per 100 individuals, significantly lower than in other European countries such as Germany, France, Italy, and the United Kingdom, where the ratio is estimated at around 5 specialists per 100 incarcerated individuals. Due to the high demand for psychological assistance and limited human resources, there is a need for brief, intensive, and evidence-based group interventions to address EDs in the penitentiary context.

Approach to Mental Health Issues in the Penitentiary System

The approach to penitentiary healthcare varies across different regions in Spain. Currently, the only autonomous communities with competencies in this area are Catalonia, the Basque Country, and the Chartered Community of Navarre. In the rest of the national territory, at the state level, this responsibility falls under the General Secretariat of Penitentiary Institutions.

Regarding strategies for the penitentiary treatment of mental health in Spain, individuals with psychological disorders who are deprived of their liberty can receive assistance through two resources: Psychiatric Penitentiary Hospitals (PPHs), institutions under the General Secretariat of Penitentiary Institutions offering treatment during incarceration, and ordinary penitentiary centers, which house 80% of inmates with mental disorders. In 2009, the Mental Illness Care Program in Prison (PAIEM) was introduced, available in 64 of the 66 ordinary centers under the Ministry of the Interior for inmates with Severe Mental Disorders. This program includes activities related to social skills promotion, self-care, improved self-control, psychoeducation, relapse prevention, and preparation for release, among others. In 2022, these interventions recorded a total of 1,817 participants, representing 4.45% of the total incarcerated population in the country.

In recent years, new models of mental health care have emerged, particularly in Catalonia, where the approach to this health issue in prisons occurs in three different areas: psychiatric units, outpatient care through the Primary Support Program (PSP), and care for individuals in third-degree through the Individualized Penitentiary Service Program (PSI). Despite these efforts, the high prevalence of mental disorders among inmates and the lack of resources significantly hinder the implementation of specific, evidence-based intervention programs.

Currently, various initiatives are being implemented to address some of the issues present in the prison population, such as self-harming behaviors. An example is the Systems Training for Emotional Predictability and Problem Solving (STEPPS) program, specifically designed to treat these behaviors. This group-based cognitive-behavioral therapeutic approach illustrates the feasibility of implementing structured group interventions in the penitentiary context.

However, given the high prevalence of EDs among inmates and the comorbidity present in these disorders, it is necessary to develop and implement transdiagnostic interventions aimed at improving emotion regulation skills across all EDs, not solely those exhibiting self-harming behaviors.

Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders and Intervention Formats

The categorical classification model of mental disorders has facilitated the development of various evidence-based psychological treatments targeting specific clinical syndromes described in the DSM or ICD manuals. Despite the benefits achieved thus far, psychopathological and clinical studies have highlighted the existence of shared etiological and maintenance mechanisms across different disorders and disorder groups, leading to the transdiagnostic approach. The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) is a manualized transdiagnostic intervention based on Cognitive Behavioral Therapy, focusing on addressing the etiological and maintenance mechanisms of EDs, such as neuroticism, worry, rumination, and emotion dysregulation, among others. The UP consists of eight modules that include training in five key emotion regulation skills: mindfulness, cognitive flexibility, counteracting emotion-driven behaviors, interoceptive exposure, and emotional exposure. Its modular nature enhances flexibility and adaptability to various clinical problems (e.g., women in fertility units or as a preventive measure for EDs in university students) and allows for cost-effective applications, such as group formats. To date, several systematic reviews and meta-analyses have supported the efficacy of the UP in treating individuals diagnosed with EDs, considering it a treatment of choice for these disorders.

In Spain, our research team has led a line of investigation focused on the evaluation, diagnosis, and treatment of EDs through the UP. In our country, the UP has proven to be an effective and cost-efficient intervention for treating EDs when applied in group format within specialized mental health units of the Public Health System. Specifically, in a multicenter randomized clinical trial involving 533 participants diagnosed with EDs, the UP was administered in 12 two-hour weekly sessions. The study's results indicated that changes in the UP treatment condition were comparable to those achieved with treatment as usual (non-structured individual cognitive-behavioral therapy), with greater improvements observed in depression, anxiety symptoms, and quality of life. Furthermore, the improvements in the UP condition were sustained over time (up to 12 months post-treatment), despite the intervention being delivered intensively over approximately three months, reflecting its long-term efficacy. Additionally, the project's findings demonstrated that, in the long term (12-month follow-up), the cost of treatment in the UP condition was lower than in the treatment-as-usual condition (€161.74, SD = 34.09, range €95.92-€299.75 vs. €183.50, SD = 77.52, range €71.94-€335.72, respectively), and high levels of participant satisfaction and strong acceptability among clinical professionals in public mental health units were also observed.

Finally, the UP has also been adapted to treat severe mental disorders, such as bipolar disorder and psychotic spectrum disorders. In the latter case, our research team has demonstrated its efficacy in individuals at high risk for psychosis. Positive outcomes have also been observed in patients with treatment-resistant schizophrenia, self-injurious behaviors, and suicidal ideation. Although some of these studies are pilot or single-case designs, the encouraging results in emotional symptoms, emotion regulation, and quality of life suggest that the UP may be a useful and complementary intervention in addressing emotional dysregulation, especially in more severe disorders. This opens up doors for further investigation into its efficacy. However, to date, no studies have examined the feasibility of the UP in the prison setting.

Study Rationale

The high prevalence of emotional disorders, along with their comorbidity with other severe mental illnesses in the prison population, presents a significant challenge due to the limited human and material resources in penitentiary centers. In this regard, the UP has proven to be an effective intervention across various contexts and emotional problems. For this reason, implementing the UP in a group format for the treatment of emotional disorders in prison settings could optimize available resources and provide a comprehensive approach to emotional disorders, improving inmates' mental health, comorbid symptomatology, and quality of life. To our knowledge, this will be the first study to test the feasibility and clinical utility of the UP for the group-based treatment of emotional disorders in prison settings, and its findings will lay the groundwork for the development of future controlled clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* At least one emotional disorder diagnosis (e.g., anxiety, depression, OCD, trauma-related, somatic, dissociative) based on the MINI interview
* Comprehension of the intervention language (Spanish or Catalan)
* Substance abstinence for more than 1 month
* Voluntary participation and availability for all assessment and treatment sessions
* Stable pharmacological treatment during the study unless medically contraindicated
* Signed informed consent

Exclusion Criteria:

* No emotional disorder diagnosis
* Cognitive impairment or IQ <70 preventing comprehension
* Diagnosis of a mental disorder incompatible with group formats (e.g., histrionic personality disorder)
* Suicide risk at assessment
* Legal status involving potential release or leave that could affect adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Structured interview for anxiety disorders and related disorders, according to the DSM-5 (ADIS-5) | Only before of the treatment to check inclusion criteria
  Diagnostic interview to determine if the participant has a clinical diagnosis of emotional disorder (ET) and can be part of the study. The following diagnoses according to the DSM-V are included within the category of emotional disorder: major depressive disorder, dysthymic disorder, panic disorder, agoraphobia, obsessive-compulsive disorder, generalized anxiety disorder, post-traumatic stress disorder, social anxiety disorder, hypochondria, and adjustment disorders. Patients with anxiety disorders not otherwise specified and those with depressive disorders not otherwise specified will also be included in the study.
General Depression Severity and Interference Scale (ODSIS) | Up to 6 months follow-up
  Severity of depressive symptoms; 5 items with 5-point Likert scale ranging from 0 (I did not feel depressed) to 4 (constant depression). Higher scores are associated with greater depressive symptomatology and interference.
General Severity and Interference Scale for Anxiety (OASIS) | Up to 6 months follow-up
  Severity of anxiety symptoms; 5 items with 5-point Likert scale ranging from 0 (I did not feel anxious) to 4 (constant anxiety). Higher scores are associated with greater anxiety symptomatology and interference.
Multidimensional Inventory for Emotional Disorders (MEDI) | Up to 6 months follow-up
  Evaluation through 49 items of the transdiagnostic profile of Emotional Disorders, which is composed of nine dimensions: neurotic temperament, positive temperament, depressed mood, somatic anxiety, arousal activation, social anxiety, intrusive cognitions, traumatic re-experiencing, and avoidance

SECONDARY OUTCOMES:
Emotional Regulation Difficulties Scale (DERS) | Up to 6 months follow-up
  The evaluation is conducted through 28 items assessing difficulties in emotional regulation, divided into 5 subscales: lack of control, rejection, interference, inattention, and emotional confusion. Scores range from 1 (almost never) to 5 (almost always), with higher scores being associated with greater difficulties in emotional regulation.
EuroQol | Up to 6 months follow-up
  Quality of life is evaluated through 5 items assessing difficulties in mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Scores range from 1 (I do not have problems) to 3 (unable to perform these activities), with higher scores being associated with a worse quality of life.
The EuroQol Visual Analog Scale (VAS) | Up to 6 months follow-up
  The EuroQol Visual Analog Scale (VAS) assesses self-reported quality of life using a thermometer scale ranging from 0 (the worst imaginable health state) to 100 (the best imaginable health state).
Satisfaction with Treatment Questionnaire (STQ) An adaptation of Client Satisfaction Questionnaire (CSQ-8) | Up to 6 months follow-up
  Our adaptation includes 6 of the 8 items of the CSQ-8 (perceived quality, adequacy to previous expectations, recommendation of the treatment to friends or family, usefulness of the techniques learned, general satisfaction with the intervention and probability that they will choose an intervention of this type again) and one more item related to the discomfort generated by the intervention. Likewise, a change has been made in the Likert response scale from 4 points in the original (0 = "Bad / Not at all" to 4 = "Excellent/Very Much") to 11 in the current one (0 = "Bad / Not at all to 10 = "Excellent/Very Much").

OTHER OUTCOMES:
Questionnaire on Sociodemographic Data (ad hoc) | Baseline
  Ad-hoc; Sex, age, marital status, number of sessions attended, and legal status of each participant.
Acceptability Questionnaire based on the TFA model | At the end of treatment (at 3 months)
  The Acceptability Questionnaire, based on the TFA model, consists of 7 items with a Likert-type response scale ranging from 1 (completely disagree, no effort, unsure, or unacceptable) to 5 (strongly agree, great effort, very sure, or completely acceptable). It evaluates the following dimensions: (1) Affective Attitude, assessing the extent to which participants liked or disliked using the UP; (2) Burden, measuring how much effort it cost to apply the UP; (3) Ethicality, evaluating whether there were any negative ethical or moral consequences of applying the UP; (4) Intervention Coherence, asking whether the approach of the UP to improve patients' emotional regulation made sense to the user; (5) Opportunity Costs, looking at whether the application of the UP interfered with other psychotherapy priorities; (6) Perceived Effectiveness, gauging how much the UP helped patients regulate their emotions; and (7) Self-efficacy, reflecting the degree of competence felt whe
Questionnaire on Intention to Use the UP in the Future and General Acceptability | At the end of treatment (at 3 months)
  The Questionnaire on Intention to Use the UP in the Future and General Acceptability includes an ad hoc question aimed at gauging participants' willingness to apply the UP again in the future. Specifically, for GHPs with experience in applying the UP, the question asks: To what extent would you accept applying it again? For participants with no prior experience, the question asks: To what extent would you accept using the UP? The response format is a 5-point Likert scale, ranging from 1 (never) to 5 (always). Higher scores are associated with greater general acceptability and a stronger intention to use the UP in the future.
Barriers to Implementation | At the end of treatment (at 3 months)
  The Barriers to Implementation Inventory (BTI) is a 39-item inventory designed to identify barriers to program implementation across four domains: equipment, administrative, theoretical/philosophical, and structural problems. Higher scores are associated with a greater number of barriers perceived during the implementation process.
Viability questionnaire (Ad hoc) | At the end of treatment (at 3 months)
  The ad-hoc questionnaire will include questions with a Likert-type scale, ranging from 0 (Not at all) to 10 (A lot), to assess therapists' opinions on aspects such as the content, exercises, format, and duration of the intervention, as well as the group dynamics and functioning. Additionally, there will be open-ended questions to allow therapists to provide more detailed and specific feedback on their experiences and perceptions, enabling a deeper and more comprehensive evaluation of the process.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Teruel, Teruel, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under request
Supporting Information: Study Protocol

REFERENCES:
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Osma J, Martinez-Loredo V, Quilez-Orden A, Peris-Baquero O, Ferreres-Galan V, Prado-Abril J, Torres-Alfosea MA, Rosellini AJ. Multidimensional emotional disorders inventory: Reliability and validity in a Spanish clinical sample. J Affect Disord. 2023 Jan 1;320:65-73. doi: 10.1016/j.jad.2022.09.140. Epub 2022 Sep 29. PMID 36183816
- [Background] Osma J, Quilez-Orden A, Suso-Ribera C, Peris-Baquero O, Norman SB, Bentley KH, Sauer-Zavala S. Psychometric properties and validation of the Spanish versions of the overall anxiety and depression severity and impairment scales. J Affect Disord. 2019 Jun 1;252:9-18. doi: 10.1016/j.jad.2019.03.063. Epub 2019 Mar 29. PMID 30953927
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Peris-Baquero O, Osma J, Gil-LaCruz M, Martinez-Garcia L. Acceptability of and intention to use the Unified Protocol delivered in group format in the Spanish Public Health System. J Eval Clin Pract. 2021 Dec;27(6):1299-1309. doi: 10.1111/jep.13546. Epub 2021 Feb 9. PMID 33565231
- [Background] Osma J, Peris-Baquero O, Suso-Ribera C, Farchione TJ, Barlow DH. Effectiveness of the Unified Protocol for transdiagnostic treatment of emotional disorders in group format in Spain: Results from a randomized controlled trial with 6-months follow-up. Psychother Res. 2022 Mar;32(3):329-342. doi: 10.1080/10503307.2021.1939190. Epub 2021 Jun 16. PMID 34132170
- [Background] Barlow DH, Harris BA, Eustis EH, Farchione TJ. The unified protocol for transdiagnostic treatment of emotional disorders. World Psychiatry. 2020 Jun;19(2):245-246. doi: 10.1002/wps.20748. No abstract available. PMID 32394551
- [Background] Sakiris N, Berle D. A systematic review and meta-analysis of the Unified Protocol as a transdiagnostic emotion regulation based intervention. Clin Psychol Rev. 2019 Aug;72:101751. doi: 10.1016/j.cpr.2019.101751. Epub 2019 Jun 25. PMID 31271848
- [Background] Cassiello-Robbins C, Southward MW, Tirpak JW, Sauer-Zavala S. A systematic review of Unified Protocol applications with adult populations: Facilitating widespread dissemination via adaptability. Clin Psychol Rev. 2020 Jun;78:101852. doi: 10.1016/j.cpr.2020.101852. Epub 2020 Apr 20. PMID 32360953
- [Background] Carlucci L, Saggino A, Balsamo M. On the efficacy of the unified protocol for transdiagnostic treatment of emotional disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Jul;87:101999. doi: 10.1016/j.cpr.2021.101999. Epub 2021 Mar 9. PMID 34098412
- See also: IPES web (Investigation group) — https://ipes-group.com/